CLINICAL TRIAL: NCT01855750
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of the Bruton's Tyrosine Kinase (BTK) Inhibitor, PCI-32765 (Ibrutinib), in Combination With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Subjects With Newly Diagnosed Non-Germinal Center B-Cell Subtype of Diffuse Large B-Cell Lymphoma
Brief Title: A Study of the Bruton's Tyrosine Kinase Inhibitor, PCI-32765 (Ibrutinib), in Combination With Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With Newly Diagnosed Non-Germinal Center B-Cell Subtype of Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR102118; PCI-32765DBL3001 (Other: Janssen Research & Development, LLC); U1111-1139-6222 (Other: Universal Trial Number); 2013-000959-40 (EudraCT Number)
Record Dates: First submitted 2013-05-14; First posted 2013-05-16 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma
Keywords: Lymphoma; B-cell lymphoma; Non-germinal center B-cell subtype; Diffuse large B-cell lymphoma; Bruton's tyrosine kinase inhibitor; PCI-32765; JNJ-54179060; Ibrutinib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone
MeSH Terms: conditions — Lymphoma; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm A: placebo + R-CHOP (Placebo Comparator): Treatment Arm A = placebo + R-CHOP (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone)
  Interventions: Drug: Placebo; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone (or equivalent)
- Treatment Arm B: ibrutinib + R-CHOP (Experimental): Treatment Arm B = ibrutinib + R-CHOP
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone (or equivalent)

INTERVENTIONS:
Drug: Ibrutinib — 560 mg capsules administered by mouth once daily (21-day cycles)
  Arms: Treatment Arm B: ibrutinib + R-CHOP
Drug: Placebo — 4 matched capsules administered by mouth once daily (21-day cycles)
  Arms: Treatment Arm A: placebo + R-CHOP
Drug: Rituximab — 375 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Cyclophosphamide — 750 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Doxorubicin — 50 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Vincristine — 1.4 mg/m2 administered intravenously once on Day 1 of each cycle (21-day cycles)
Drug: Prednisone (or equivalent) — 100 mg capsules administered by mouth once daily on Day 1 to Day 5 of each cycle

SUMMARY:
The purpose of this study is to evaluate if ibrutinib administered in combination with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) improves the clinical outcome in newly diagnosed patients with non-germinal center B-cell subtype (GCB) of diffuse large B-cell lymphoma (DLBCL) selected by immunohistochemistry (IHC) or newly diagnosed patients with activated B cell-like (ABC) subtype of DLBCL identified by gene expression profiling (GEP) or both populations.

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), double-blind (individuals and study personnel will not know the identity of study treatments), placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial)-controlled study to compare the efficacy and safety of ibrutinib in combination with R-CHOP versus R-CHOP alone in adult patients newly diagnosed non-GCB DLBCL selected by IHC or newly diagnosed patients with ABC subtype of DLBCL identified by GEP or both populations. The study will include screening, active treatment, and posttreatment follow-up phases. The study will end when 50% of participants have died or 5 years after the last participant is randomized or the sponsor terminates the study, whichever occurs first. Approximately 800 participants will be randomly assigned in a 1:1 ratio to receive either placebo+R-CHOP (treatment arm A) or ibrutinib+R-CHOP (treatment arm B). All participants will receive R-CHOP as background therapy for 6 or 8 cycles (21 days per cycle) prespecified according to local practice. After 4 treatment cycles, an interim response assessment will be performed to evaluate disease progression for each participant. Participants with progressive disease or relapsed disease after complete response will be discontinued from treatment. Participants who discontinue R-CHOP without disease progression will continue study drug (placebo or ibrutinib) until 6 or 8 cycles are completed, disease progression, or unacceptable toxicity, whichever occurs first. After completion of study drug, participants will undergo assessment of tumor response based on the Revised Response Criteria for Malignant Lymphoma. Participants with documented residual disease upon completion of at least 6 cycles of R-CHOP therapy are considered eligible to initiate subsequent antilymphoma therapy. Serial pharmacokinetic samples will be collected before and after dosing, and safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* No prior treatment for diffuse B-cell lymphoma (DLBCL)
* Histologically-confirmed non-germinal center B-cell subtype DLBCL
* Stage II (not candidates for local x-ray therapy), III, or IV disease by the Ann Arbor Classification
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma
* Revised International Prognostic Index score of >=1
* Eastern Cooperative Oncology Group performance status grade of 0, 1, or 2
* Hematology and biochemical laboratory values within protocol-defined parameters prior to random assignment and at baseline
* Left ventricular ejection fraction within institutional normal limits, as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan
* Agrees to protocol-defined use of effective contraception (for women, these restrictions apply for 12 months after the last dose of rituximab or 1 month after the last dose of study drug, whichever is later; for men, these restrictions apply for 12 months after the last dose of rituximab or 3 months after the last dose of study drug, whichever is later)
* Men must agree to not donate sperm during and after the study for 12 months after the last dose of rituximab or 3 months after the last dose of study drug, whichever is later
* Women of childbearing potential must have a negative serum or urine pregnancy test at screening

Exclusion Criteria:

* Major surgery within 4 weeks of random assignment
* Known central nervous system or primary mediastinal lymphoma
* Prior history of indolent lymphoma
* Diagnosed or treated for malignancy other than DLBCL, except: malignancy treated with curative intent and with no known active disease present for >=3 years before random assignment; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma in situ without evidence of disease
* History of stroke or intracranial hemorrhage within 6 months prior to random assignment
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors
* Prior anthracycline use >=150 mg/m2
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of human immunodeficiency virus or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous antibiotics
* Women who are pregnant or breastfeeding
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 838 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2019-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (201):
- United States (44):
  - Tucson, Arizona
  - Greenbrae, California
  - La Jolla, California
  - Los Angeles, California
  - Salinas, California
  - Stanford, California
  - Danbury, Connecticut
  - Hartford, Connecticut
  - Washington D.C., District of Columbia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Peoria, Illinois
  - Fort Wayne, Indiana
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Topeka, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Omaha, Nebraska
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - Fresh Meadows, New York
  - Johnson City, New York
  - Mineola, New York
  - New York, New York
  - Rochester, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - North Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Temple, Texas
  - Burlington, Vermont
  - Seattle, Washington
- Argentina (2):
  - Buenos Aires
  - Ciudad de Buenos Aires
- Australia (10):
  - Adelaide
  - Concord
  - Darlinghurst
  - Hobart
  - Melbourne
  - Nedlands
  - Perth
  - Randwick
  - South Brisbane
  - Woolloongabba
- Belgium (7):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Haine Saint Paul La Louviere
  - Kortrijk
  - Leuven
- Brazil (3):
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Toronto, Ontario
  - Lévis, Quebec
  - Montreal, Quebec
- China (10):
  - Beijing
  - Changchun
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Harbin
  - Jinan
  - Nanjing
  - Shanghai
  - Tianjin
- Czechia (4):
  - Brno
  - Hradec Králové
  - Ostrava
  - Prague
- Denmark (4):
  - Aarhus N
  - Copenhagen
  - Roskilde
  - Vejle
- Finland (4):
  - Helsinki
  - Jyväskylä
  - Oulu
  - Turku
- France (8):
  - Grenoble
  - Limoges
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rouen
  - Tours
  - Villejuif
- Germany (10):
  - Augsburg
  - Bamberg
  - Berlin
  - Dresden
  - Essen
  - Frankfurt
  - Jena
  - München
  - Münster
  - Villingen-Schwenningen
- Hungary (5):
  - Budapest
  - Debrecen
  - Gyula
  - Szombathely
  - Veszprém
- Israel (6):
  - Beersheba
  - Hadera
  - Haifa
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Japan (17):
  - Fukuoka
  - Hiroshima
  - Isehara
  - Kobe
  - Kumamoto
  - Kyoto
  - Nagano
  - Nagoya
  - Narita
  - Osaka
  - Ōsaka-sayama
  - Sapporo
  - Sendai
  - Suita
  - Tachikawa
  - Tokyo
  - Tsukuba
- Mexico (3):
  - México
  - Monterrey
  - San Luis Potosí City
- Netherlands (7):
  - Amsterdam-Zuidoost
  - Arnhem
  - Dordrecht
  - Groningen
  - Leiden
  - Nieuwegein
  - Rotterdam
- Norway (2):
  - Oslo
  - Tromsø
- Poland (8):
  - Brzozów
  - Chorzów
  - Krakow
  - Lodz
  - Olsztyn
  - Poznan
  - Warsaw
  - Wroclaw
- Russia (7):
  - Moscow
  - Nizhny Novgorod
  - Rostov-on-Don
  - Saint Petersburg
  - Sochi
  - Volgograd
  - Yekaterinburg
- South Korea (3):
  - Busan
  - Goyang-si
  - Seoul
- Spain (4):
  - Barcelona
  - Madrid
  - Salamanca
  - Seville
- Sweden (4):
  - Linköping
  - Luleå
  - Lund
  - Uppsala
- Taiwan (3):
  - Taichung
  - Tainan
  - Taoyuan
- Turkey (Türkiye) (6):
  - Adana
  - Ankara
  - Istanbul
  - Izmir
  - Kayseri
  - Samsun
- Ukraine (5):
  - Cherkassy
  - Khmelnitskiy
  - Kiev
  - Lviv
  - Makiivka
- United Kingdom (9):
  - Glasgow
  - Liverpool
  - London
  - Maidstone
  - Manchester
  - Nottingham
  - Oxford
  - Romford
  - Southampton

REFERENCES:
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Johnson PWM, Balasubramanian S, Hodkinson B, Shreeve SM, Sun S, Srinivasan S, Steele AJ, Vermeulen J, Sehn LH, Wilson WH. Clinical impact of ibrutinib plus R-CHOP in untreated DLBCL coexpressing BCL2 and MYC in the phase 3 PHOENIX trial. Blood Adv. 2023 May 23;7(10):2008-2017. doi: 10.1182/bloodadvances.2022009389. PMID 36696540
- [Derived] Wilson WH, Wright GW, Huang DW, Hodkinson B, Balasubramanian S, Fan Y, Vermeulen J, Shreeve M, Staudt LM. Effect of ibrutinib with R-CHOP chemotherapy in genetic subtypes of DLBCL. Cancer Cell. 2021 Dec 13;39(12):1643-1653.e3. doi: 10.1016/j.ccell.2021.10.006. Epub 2021 Nov 4. PMID 34739844
- [Derived] Younes A, Sehn LH, Johnson P, Zinzani PL, Hong X, Zhu J, Patti C, Belada D, Samoilova O, Suh C, Leppa S, Rai S, Turgut M, Jurczak W, Cheung MC, Gurion R, Yeh SP, Lopez-Hernandez A, Duhrsen U, Thieblemont C, Chiattone CS, Balasubramanian S, Carey J, Liu G, Shreeve SM, Sun S, Zhuang SH, Vermeulen J, Staudt LM, Wilson W; PHOENIX investigators. Randomized Phase III Trial of Ibrutinib and Rituximab Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Non-Germinal Center B-Cell Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2019 May 20;37(15):1285-1295. doi: 10.1200/JCO.18.02403. Epub 2019 Mar 22. PMID 30901302

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm B: Ibrutinib+R-CHOP: Participants received ibrutinib 560 milligram (mg) (4*140 mg) capsules orally once daily (Cycle 1 Day 1 to Day 21 of last cycle; 21-day cycles) along with R-CHOP (Rituximab - Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone) as a background chemotherapy. R-CHOP regimen included rituximab 375 milligram per square meter (mg/m^2) intravenously (IV), cyclophosphamide 750 mg/m^2 IV, doxorubicin 50 mg/m^2 IV, and vincristine 1.4 mg/m^2 IV, administered on Day 1 and prednisone 100 mg capsules orally on Days 1 to 5 of each cycle. Participants received background chemotherapy plus ibrutinib for 6 or 8 cycles per site preference (21 days per cycle).
- Treatment Arm A: Placebo+R-CHOP: Participants received matching placebo (4 capsules) orally once daily (21-day cycles) along with R-CHOP background chemotherapy. R-CHOP regimen included rituximab 375 milligram per square meter (mg/m^2) intravenously (IV), cyclophosphamide 750 mg/m^2 IV, doxorubicin 50 mg/m^2 IV, and vincristine 1.4 mg/m^2 IV, administered on Day 1 and prednisone 100 mg capsules orally on Days 1 to 5 of each cycle. Participants received background chemotherapy plus matching placebo for 6 or 8 cycles per site preference (21 days per cycle).
Period: Overall Study
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Started | 419 | 419
Treated | 416 (3 participants not treated:2 withdrew consent and 1 not treated per Sponsor/investigator's decision.) | 418 (1 participant not treated: withdrew consent.)
Completed | 0 | 0
Not Completed | 419 | 419
Not completed — Death | 78 | 78
Not completed — Lost to Follow-up | 9 | 23
Not completed — Withdrawal by Subject | 35 | 28
Not completed — Sponsor ends the study | 297 | 290

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP | Total
Number analyzed (Participants) | 419 | 419 | 838
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (12.57) | 58.8 (13.57) | 59.9 (13.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 193 | 391
  Male | 221 | 226 | 447
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 13 | 30
  Not Hispanic or Latino | 388 | 396 | 784
  Unknown or Not Reported | 14 | 10 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 237 | 250 | 487
  Black or African American | 4 | 4 | 8
  Asian | 166 | 160 | 326
  American Indian or Alaska Native | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 1 | 2
  Unknown | 0 | 0 | 0
  Not reported | 7 | 2 | 9
  Multiple | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 1 | 2
  Australia | 12 | 8 | 20
  Belgium | 8 | 7 | 15
  Brazil | 8 | 4 | 12
  Canada | 12 | 9 | 21
  China | 104 | 96 | 200
  Czech Republic | 18 | 12 | 30
  Denmark | 5 | 6 | 11
  Finland | 6 | 8 | 14
  France | 7 | 4 | 11
  Germany | 5 | 8 | 13
  Hungary | 5 | 6 | 11
  Israel | 11 | 12 | 23
  Italy | 24 | 18 | 42
  Japan | 33 | 40 | 73
  Mexico | 2 | 1 | 3
  Netherlands | 5 | 1 | 6
  Norway | 1 | 6 | 7
  Poland | 15 | 24 | 39
  Russia | 19 | 34 | 53
  Korea, Republic Of | 14 | 11 | 25
  Spain | 5 | 7 | 12
  Sweden | 0 | 1 | 1
  Taiwan, Province Of China | 8 | 9 | 17
  Turkey | 27 | 24 | 51
  Ukraine | 10 | 9 | 19
  United Kingdom | 14 | 17 | 31
  United States | 40 | 36 | 76

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS) - Intent-to-Treat (ITT) Population
Description: EFS: duration from randomization date to disease progression(PD) date, relapse from complete response(CR) assessed by investigator, initiation of subsequent systemic antilymphoma therapy for either positron emission tomography(PET)-positive/ biopsy-proven residual disease upon completion of >=6 cycles of R-CHOP therapy/death, whichever occurred first. Responses were based on Revised Response Criteria for Malignant Lymphoma. PD: any new lesion or increase by 50% of previously involved sites from nadir; PD criteria: Appearance of new nodal lesion 1.5 cm in any axis, 50% increase in sum of product of diameters(SPD) of >1 node or 50% increase in longest diameter of previously identified node 1 cm in short axis. CR: disappearance of all evidence of disease; CR criteria: nodal masses PET positive prior to therapy; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy.
Time Frame: Up to 5.5 years
Population: Intent-to-Treat (ITT) population included all randomized participants, enrolled with non-germinal center B-cell (GCB) of diffuse large B-cell lymphoma (DLBCL) subtype by immunohistochemistry (IHC), and were analyzed according to treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Number analyzed (Participants) | 419 | 419
Months | 49.64 [47.47 to NA] — Here NA signifies that the upper limit of Confidence Interval (CI) was not estimable due to lesser number of events. | 54.77 [48.16 to 54.77]
Statistical Analysis 1: Comparison: Treatment Arm B: Ibrutinib+R-CHOP vs Treatment Arm A: Placebo+R-CHOP; Test type: Superiority; p = 0.5167, Log Rank; Hazard Ratio (HR) = 0.922, 95% CI 2-sided [0.720 to 1.180]

2. Primary Outcome: Event-Free Survival (EFS) - Activated B-Cell (ABC) Population
Description: EFS: duration from randomization date to PD date, relapse from CR assessed by investigator, initiation of subsequent systemic antilymphoma therapy for either PET-positive/ biopsy-proven residual disease upon completion of >=6 cycles of R-CHOP therapy/death, whichever occurred first. Responses were based on Revised Response Criteria for Malignant Lymphoma. PD: any new lesion or increase by 50% of previously involved sites from nadir; PD criteria: Appearance of new nodal lesion 1.5 cm in any axis, 50% increase in SPD of >1 node or 50% increase in longest diameter of previously identified node 1 cm in short axis. CR: disappearance of all evidence of disease; CR criteria: nodal masses PET positive prior to therapy; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy.
Time Frame: Up to approximately 4.5 years
Population: ABC population included ITT population (all randomized participants, enrolled with non-GCB of DLBCL subtype by IHC) having ABC subtype determined by gene expression profiling (GEP) (retrospectively determined from available formalin-fixed paraffin-embedded [FFPE] tissue specimens). Participants were analyzed according to randomized treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Number analyzed (Participants) | 285 | 282
Months | 48.56 [48.56 to NA] — Here NA signifies that the upper limit of CI was not estimable due to lesser number of events. | 48.16 [48.16 to NA] — Here NA signifies that the upper limit of CI was not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Treatment Arm B: Ibrutinib+R-CHOP vs Treatment Arm A: Placebo+R-CHOP; Test type: Superiority; p = 0.7311, Log Rank; Hazard Ratio (HR) = 0.949, 95% CI 2-sided [0.704 to 1.279]

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the duration from the date of randomization to the date of progression, relapse from CR, or death, whichever occurred first. Responses were based on Revised Response Criteria for Malignant Lymphoma. Progressive Disease (PD): any new lesion or increase by 50% of previously involved sites from nadir; PD criteria: Appearance of new nodal lesion 1.5 centimeter (cm) in any axis, 50% increase in SPD of >1 node or 50% increase in longest diameter of previously identified node 1 cm in short axis. CR: disappearance of all evidence of disease; CR criteria: nodal masses PET positive prior to therapy; mass of any size permitted if PET negative; regression to normal size on CT; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy.
Time Frame: Up to approximately 4.5 years
Population: ITT population included all randomized participants, enrolled with non-GCB of DLBCL subtype by IHC, and were analyzed according to treatment to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Number analyzed (Participants) | 419 | 419
Months | 48.56 [48.56 to NA] — Here NA signifies that the upper limit of Confidence Interval (CI) was not estimable due to lesser number of events. | NA [48.16 to NA] — Here NA signifies that median and the upper limit of Confidence Interval (CI) were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Treatment Arm B: Ibrutinib+R-CHOP vs Treatment Arm A: Placebo+R-CHOP; Test type: Superiority; p = 0.5027, Log Rank; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.710 to 1.183]

4. Secondary Outcome: Percentage of Participants Who Achieved Complete Response (CR)
Description: Percentage of participants with measurable disease who achieved CR were reported. CR: disappearance of all evidence of disease. CR Criteria: Complete disappearance of all disease-related symptoms; all lymph nodes and nodal masses regressed to normal size (less than or equal to [<=]1.5 cm in greatest transverse diameter [GTD] for nodes greater than [>]1.5 cm before therapy). Previous nodes of 1.1 to 1.5 cm in long axis and greater than (>)1.0 cm in short axis before treatment decreased to <=1.0 cm in short axis after treatment. Disappearance of all splenic and hepatic nodules and other extranodal disease; a negative positron emission tomography (PET) scan. A posttreatment residual mass of any size but PET-negative; spleen and liver: not palpable, nodules disappeared; bone marrow: infiltrate cleared on repeat biopsy.
Time Frame: Up to approximately 4.5 years
Population: ITT population included all randomized participants, who were enrolled with the non-GCB of DLBCL subtype by IHC. Participants in this population were analyzed according to the treatment to which they were randomized.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Number analyzed (Participants) | 419 | 419
Percentage of participants | 67.3 | 68.0
Statistical Analysis 1: Comparison: Treatment Arm B: Ibrutinib+R-CHOP vs Treatment Arm A: Placebo+R-CHOP; Test type: Superiority; p = 0.8229, Cochran-Mantel-Haenszel (CMH) Chi-square; Odds Ratio (OR) = 0.967, 95% CI 2-sided [0.722 to 1.296]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the duration from the date of randomization to the date of the participant's death. Median Overall Survival was estimated by using the Kaplan-Meier method.
Time Frame: Up to 5.5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Number analyzed (Participants) | 419 | 419
Months | NA [NA to NA] — Here NA signifies that the median, lower and upper limit of CI were not estimable due to lesser number of events. | NA [NA to NA] — Here NA signifies that the median, lower and upper limit of CI were not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Treatment Arm B: Ibrutinib+R-CHOP vs Treatment Arm A: Placebo+R-CHOP; Test type: Superiority; p = 0.8549, Log Rank; Hazard Ratio (HR) = 1.030, 95% CI 2-sided [0.754 to 1.407]

6. Secondary Outcome: Time to Worsening in the Lymphoma Subscale of Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym)
Description: Time to worsening in the Lymphoma subscale of the FACT-Lym, defined as the interval from the date of randomization to the start date of worsening of participant symptoms. Worsening was defined by a 5-point decrease from baseline. FACT-Lym Lymphoma subscale contains 15 questions, scores from 0 to 4 for each question (higher the worse). Lymphoma subscale score is the total of reverse scores, range 0 to 60. Higher scores indicate a better quality of life.
Time Frame: Up to approximately 4.5 years
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
Number analyzed (Participants) | 419 | 419
Months | 11.7 [4.9 to 23.5] | 35.0 [19.8 to NA] — Here NA signifies that the upper limit of CI was not estimable due to lesser number of events.
Statistical Analysis 1: Comparison: Treatment Arm B: Ibrutinib+R-CHOP vs Treatment Arm A: Placebo+R-CHOP; Test type: Superiority; p = 0.0021, Log Rank; Hazard Ratio (HR) = 1.358, 95% CI 2-sided [1.115 to 1.654]

ADVERSE EVENTS:
Time Frame: Up to 5.5 years
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Treatment Arm B: Ibrutinib+R-CHOP | Treatment Arm A: Placebo+R-CHOP
All-Cause Mortality (participants affected / at risk) | 78/416 | 78/418
Serious Adverse Events (participants affected / at risk) | 221/416 | 143/418
Other Adverse Events (participants affected / at risk) | 411/416 | 411/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm B: Ibrutinib+R-CHOP (N=416) | Treatment Arm A: Placebo+R-CHOP (N=418)
Anaemia (Blood and lymphatic system disorders) | 15 | 5
Febrile Neutropenia (Blood and lymphatic system disorders) | 78 | 44
Leukopenia (Blood and lymphatic system disorders) | 4 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 17 | 13
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 1
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 2 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 13 | 2
Atrial Flutter (Cardiac disorders) | 1 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 2 | 5
Cardiac Failure Acute (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1
Myocardial Ischaemia (Cardiac disorders) | 2 | 0
Sinus Node Dysfunction (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0
Congenital Neuropathy (Congenital, familial and genetic disorders) | 0 | 1
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Eye Haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 15 | 4
Diverticular Perforation (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric Haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastric Perforation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 2 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Mechanical Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 3
Neutropenic Colitis (Gastrointestinal disorders) | 1 | 0
Obstruction Gastric (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Small Intestinal Perforation (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 8 | 2
Asthenia (General disorders) | 2 | 1
Chest Pain (General disorders) | 1 | 0
Device Related Thrombosis (General disorders) | 0 | 1
Drowning (General disorders) | 0 | 1
Fatigue (General disorders) | 5 | 1
General Physical Health Deterioration (General disorders) | 2 | 1
Injection Site Extravasation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal Inflammation (General disorders) | 3 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 12 | 11
Sudden Death (General disorders) | 2 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 2 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 2
Arteritis Infective (Infections and infestations) | 1 | 0
Aspergillus Infection (Infections and infestations) | 2 | 0
Atypical Pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Brain Abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cerebral Aspergillosis (Infections and infestations) | 1 | 0
Clostridial Infection (Infections and infestations) | 2 | 0
Cryptococcal Fungaemia (Infections and infestations) | 1 | 0
Cytomegalovirus Gastrointestinal Infection (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 4 | 1
Enterococcal Sepsis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis Bacterial (Infections and infestations) | 0 | 1
Haemophilus Infection (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 1
Hepatitis B Reactivation (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 2 | 3
Incision Site Infection (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 2
Klebsiella Sepsis (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection Fungal (Infections and infestations) | 1 | 0
Lung Abscess (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 14 | 7
Lymph Gland Infection (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 1 | 0
Neutropenic Infection (Infections and infestations) | 2 | 1
Neutropenic Sepsis (Infections and infestations) | 1 | 2
Peritonitis (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 28 | 14
Pneumonia Cryptococcal (Infections and infestations) | 1 | 0
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia Klebsiella (Infections and infestations) | 2 | 0
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 | 1
Pseudomembranous Colitis (Infections and infestations) | 1 | 0
Pulmonary Mycosis (Infections and infestations) | 1 | 0
Respiratory Syncytial Virus Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection Bacterial (Infections and infestations) | 1 | 0
Respiratory Tract Infection Fungal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 3
Septic Shock (Infections and infestations) | 5 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 1
Urinary Tract Infection (Infections and infestations) | 5 | 3
Urosepsis (Infections and infestations) | 1 | 1
Viral Infection (Infections and infestations) | 2 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Wound Infection (Infections and infestations) | 0 | 1
Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 2
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Pubis Fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull Fractured Base (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 3
Alanine Aminotransferase Increased (Investigations) | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 5 | 2
Platelet Count Decreased (Investigations) | 2 | 0
Weight Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 3 | 0
White Blood Cell Count Increased (Investigations) | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 8 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis Pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Angioimmunoblastic T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered State of Consciousness (Nervous system disorders) | 1 | 0
Central Nervous System Inflammation (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 | 1
Cerebrovascular Disorder (Nervous system disorders) | 1 | 0
Dizziness Postural (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Febrile Convulsion (Nervous system disorders) | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 2 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Intracranial Hypotension (Nervous system disorders) | 0 | 1
Nerve Compression (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 5 | 1
Bipolar I Disorder (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 4 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 2
Urinary Retention (Renal and urinary disorders) | 1 | 0
Vaginal Fistula (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diffuse Alveolar Damage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Obliterative Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Sinus Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 2
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 6 | 1
Shock Haemorrhagic (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Vena Cava Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm B: Ibrutinib+R-CHOP (N=416) | Treatment Arm A: Placebo+R-CHOP (N=418)
Anaemia (Blood and lymphatic system disorders) | 173 | 116
Febrile Neutropenia (Blood and lymphatic system disorders) | 41 | 22
Leukopenia (Blood and lymphatic system disorders) | 70 | 74
Lymphopenia (Blood and lymphatic system disorders) | 23 | 36
Neutropenia (Blood and lymphatic system disorders) | 213 | 248
Thrombocytopenia (Blood and lymphatic system disorders) | 102 | 53
Abdominal Pain (Gastrointestinal disorders) | 37 | 34
Abdominal Pain Upper (Gastrointestinal disorders) | 28 | 34
Constipation (Gastrointestinal disorders) | 111 | 110
Diarrhoea (Gastrointestinal disorders) | 149 | 81
Dry Mouth (Gastrointestinal disorders) | 22 | 17
Dyspepsia (Gastrointestinal disorders) | 26 | 22
Mouth Ulceration (Gastrointestinal disorders) | 32 | 20
Nausea (Gastrointestinal disorders) | 170 | 135
Stomatitis (Gastrointestinal disorders) | 64 | 47
Vomiting (Gastrointestinal disorders) | 91 | 59
Asthenia (General disorders) | 28 | 16
Fatigue (General disorders) | 138 | 102
Malaise (General disorders) | 25 | 21
Mucosal Inflammation (General disorders) | 34 | 23
Oedema Peripheral (General disorders) | 46 | 29
Pyrexia (General disorders) | 83 | 68
Pneumonia (Infections and infestations) | 22 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 35 | 29
Urinary Tract Infection (Infections and infestations) | 24 | 15
Infusion Related Reaction (Injury, poisoning and procedural complications) | 23 | 26
Alanine Aminotransferase Increased (Investigations) | 25 | 24
Lymphocyte Count Decreased (Investigations) | 44 | 42
Neutrophil Count Decreased (Investigations) | 99 | 81
Platelet Count Decreased (Investigations) | 83 | 38
Weight Decreased (Investigations) | 36 | 18
White Blood Cell Count Decreased (Investigations) | 107 | 104
Decreased Appetite (Metabolism and nutrition disorders) | 64 | 51
Hypoalbuminaemia (Metabolism and nutrition disorders) | 24 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 75 | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 22 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 28 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 34 | 40
Bone Pain (Musculoskeletal and connective tissue disorders) | 17 | 21
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 30 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 24
Dysgeusia (Nervous system disorders) | 26 | 19
Headache (Nervous system disorders) | 29 | 43
Hypoaesthesia (Nervous system disorders) | 28 | 22
Neuropathy Peripheral (Nervous system disorders) | 65 | 35
Paraesthesia (Nervous system disorders) | 28 | 16
Peripheral Sensory Neuropathy (Nervous system disorders) | 77 | 63
Insomnia (Psychiatric disorders) | 39 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 25
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 32 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 69 | 106
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 21
Rash (Skin and subcutaneous tissue disorders) | 22 | 21
Hypertension (Vascular disorders) | 23 | 18
Hypotension (Vascular disorders) | 23 | 10

LIMITATIONS AND CAVEATS:
Sponsor decided to stop the study as all participants had concluded study treatment and outcomes were not expected to change and study was considered as completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/50/NCT01855750/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT01855750/SAP_001.pdf